CLINICAL TRIAL: NCT00535730
Title: A Phase III Double-Blind, Randomized, Multicenter Study to Evaluate the Safety, Tolerability, and Immunogenicity of ZOSTAVAX™ Administered Concomitantly Versus Nonconcomitantly With PNEUMOVAX™ 23 in Subjects 60 Years of Age and Older
Brief Title: ZOSTAVAX™ Administered Concomitantly With PNEUMOVAX™ 23 (V211-012)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-012; 2007_592
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Results first posted 2009-05-13 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Herpes Zoster; Pneumococcal Infection
MeSH Terms: conditions — Herpes Zoster; Pneumococcal Infections | interventions — Herpes Zoster Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator): Placebo Comparator
  Interventions: Biological: Zoster Vaccine, Live, (Oka-Merck), ZOSTAVAX™; Biological: Comparator: placebo (concomitant-vaccine matched)
- 2 (Experimental): vaccine
  Interventions: Biological: Zoster Vaccine, Live, (Oka-Merck), ZOSTAVAX™; Biological: Pneumococcal Vaccine, Polyvalent (23-valent), PNEUMOVAX™ 23

INTERVENTIONS:
Biological: Zoster Vaccine, Live, (Oka-Merck), ZOSTAVAX™ — 0.65 mL injection Zoster Vaccine, Live, (Oka-Merck) over 4 week vaccination period
  Other Names: ZOSTAVAX™
Biological: Comparator: placebo (concomitant-vaccine matched) — Pneumococcal Vaccine, Polyvalent (23-valent) 0.5 mL Placebo injection over 4 week vaccination period.
  Arms: 1
Biological: Pneumococcal Vaccine, Polyvalent (23-valent), PNEUMOVAX™ 23 — Pneumococcal Vaccine, Polyvalent (23-valent) 0.5 mL injection over 4 week vaccination period.
  Other Names: PNEUMOVAX™ 23
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Zoster Vaccine Live and Pneumococcal Vaccine, polyvalent are as well tolerated and immunogenic when the vaccines are given together (in different body sites), as when they are given alone, in adults 60 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Stable underlying conditions
* Postmenopausal if female
* Afebrile

Exclusion Criteria:

* Previously vaccinated with either vaccine
* Immune deficiency
* History of allergy to components in either vaccine
* Concomitant antiviral therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] MacIntyre CR, Egerton T, McCaughey M, Parrino J, Campbell BV, Su SC, Pagnoni MF, Stek JE, Xu J, Annunziato PW, Chan IS, Silber JL. Concomitant administration of zoster and pneumococcal vaccines in adults >/=60 years old. Hum Vaccin. 2010 Nov;6(11):894-902. doi: 10.4161/hv.6.11.12852. Epub 2010 Nov 1. PMID 20980796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First subject enrolled on 18-Jun-2007.
  Last subject enrolled on 05-Dec-2007.
  The last subject's last visit was 11-Feb-2008.
  The study was conducted at 18 study centers throughout Canada, Australia, and Europe.
Groups:
- Nonconcomitant Group: Subjects were administered PNEUMOVAX™ 23 intramuscularly on Day 1 followed by ZOSTAVAX™ subcutaneously on Week 4
- Concomitant Group: Subjects were administered ZOSTAVAX™ subcutaneously concomitantly with PNEUMOVAX™ 23 intramuscularly at separate injection sites at Day 1
Period: Overall Study
Arm/Group | Nonconcomitant Group | Concomitant Group
Started | 236 | 237 (Two subjects were allocated but not vaccinated making the number of subjects vaccinated 235)
Completed | 234 | 230
Not Completed | 2 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nonconcomitant Group | Concomitant Group | Total
Number analyzed (Participants) | 236 | 235 | 471
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (5.6) | 66.3 (5.6) | 66.2 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 138 | 273
  Male | 101 | 97 | 198
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 2
  Black or African American | 0 | 1 | 1
  White | 235 | 233 | 468

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Varicella-zoster Virus (VZV) Antibody Responses at 4 Weeks Postvaccination
Description: GMT of the VZV antibody responses at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 and those who receive ZOSTAVAX™ and PNEUMOVAX™ 23 nonconcomitantly.
  *gpELISA = glycoprotein enzyme-linked immunosorbent assay
Time Frame: 4 weeks postvaccination
Population: Analysis was per protocol. The following protocol violations resulted in exclusion of subjects from analysis: receipt of prohibited medications; vaccine temperature compromised prior to administration; excluded medical condition; samples collected outside of Statistical Analysis Plan specified time window; exposure to herpes zoster (HZ) or VZV.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units*/mL
Arm/Group | Nonconcomitant Group | Concomitant Group
Number analyzed (Participants) | 225 | 217
gpELISA units*/mL | 448.5 [400.3 to 502.4] | 371.6 [328.7 to 420.0]
Statistical Analysis 1: Comparison: Nonconcomitant Group vs Concomitant Group; The hypothesis was that the GMT of the VZV antibody responses at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 will be noninferior to that in subjects who receive ZOSTAVAX™ nonconcomitantly; Test type: Non-Inferiority or Equivalence — The power for the noninferiority hypothesis of VZV antibody titers is 92%. The noninferiority margin is the lower bound of the two-sided 95% confidence interval on the VZV antibody GMT ratio[concomitant/nonconcomitant] being >0.67; p = 0.244, longitudinal regression model — The threshold for statistical significance is 0.025. There is no adjustment for multiple comparisons; Week 4 postvac, estimated responses, GMT ratio, 95% CI, p-value based on a longitudinal regression model adjusting for prevac titers and age (years)

2. Secondary Outcome: Safety and Tolerability of Both Vaccines When Administered Concomitantly.
Description: All adverse events were analyzed including serious adverse events; injection-site adverse events; Vaccination Report Card prompted systemic adverse events, including varicella-like rashes or herpes zoster-like rashes; all other systemic adverse events.
Time Frame: Eight weeks postvaccination
Population: All subjects who received at least one vaccination
Measure: Number; unit: Participants
Arm/Group | Nonconcomitant Group | Concomitant Group
Number analyzed (Participants) | 236 | 235
Participants
  Injection site AEs | 141 | 136
  Systemic AEs | 74 | 70
  Serious AEs | 4 | 2
  Varicella-like Rash | 3 | 2
  Zoster-like Rash | 1 | 1

3. Primary Outcome: Geometric Mean Fold Rise (GMFR) of the Varicella-zoster Virus (VZV) Antibody Responses From Day 1 to 4 Weeks Postvaccination.
Description: GMFR of the VZV antibody response from prevaccination to Week 4 postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23.
  gpELISA = glycoprotein enzyme-linked immunosorbent assay.
Time Frame: Four weeks postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Concomitant Group
Number analyzed (Participants) | 217
gpELISA units/mL | 1.9 [1.7 to 2.1]
Statistical Analysis 1: Comparison: Concomitant Group; The hypothesis was that ZOSTAVAX™ elicits an acceptable VZV antibody response when administered concomitantly with PNEUMOVAX™ 23; Test type: Superiority or Other; p < 0.001, t-test, 1 sided — The threshold for statistical significance is 0.025. There is no adjustment for multiple comparisons; The one-sided p-value for testing acceptability for GMFR is computed based on t-test. CI is computed based on the t distribution

4. Primary Outcome: Geometric Mean Titer (GMT) of the Pneumococcal Polysaccharide (PnPs) Serotype 3 Antibody Response at 4 Weeks Postvaccination.
Description: GMT of the PnPs serotype 3 antibody response at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 and those who receive ZOSTAVAX™ and PNEUMOVAX™ 23 nonconcomitantly.
Time Frame: Four weeks postvaccination
Population: Analysis was per protocol. The following protocol violations resulted in exclusion of subjects from analysis: prior receipt of a pneumococcal vaccine; receipt of prohibited medications; vaccine temperature compromised prior to administration; excluded medical condition; samples collected outside of Statistical Analysis Plan specified time window.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/mL
Arm/Group | Nonconcomitant Group | Concomitant Group
Number analyzed (Participants) | 228 | 219
micrograms/mL | 1.2 [1.1 to 1.4] | 1.1 [1.0 to 1.2]
Statistical Analysis 1: Comparison: Nonconcomitant Group vs Concomitant Group; The hypothesis was that the GMT of the PnPs antibody response to serotype 3 at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 will be noninferior to those in subjects who receive ZOSTAVAX™ nonconcomitantly; Test type: Non-Inferiority or Equivalence — The power for the noninferiority hypothesis regarding PnPs antibody titer is ~99%. The noninferiority margin is the lower bound of the two-sided 95% confidence interval (CI) on the PnPs antibody GMT ratio [concomitant/nonconcomitant] being >05; p < 0.001, longitudinal regression model — The threshold for statistical significance is 0.025. There is no adjustment for multiple comparisons; [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: Geometric Mean Titer (GMT) of the Pneumococcal Polysaccharide (PnPs) Serotype 14 Antibody Response at 4 Weeks Postvaccination.
Description: GMT of the PnPs serotype 14 antibody response at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 and those who receive ZOSTAVAX™ and PNEUMOVAX™ 23 nonconcomitantly.
Time Frame: Four weeks postvaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/mL
Arm/Group | Nonconcomitant Group | Concomitant Group
Number analyzed (Participants) | 228 | 219
micrograms/mL | 26.5 [22.9 to 30.8] | 25.7 [21.8 to 30.3]
Statistical Analysis 1: Comparison: Nonconcomitant Group vs Concomitant Group; The hypothesis was that the GMT of the PnPs antibody responses to serotype 14 at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 will be noninferior to those in subjects who receive ZOSTAVAX™ nonconcomitantly; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, longitudinal regression model — The threshold for statistical significance is 0.025. There is no adjustment for multiple comparisons; [statistical method as in outcome 1, analysis 1]

6. Primary Outcome: Geometric Mean Titer (GMT) of the Pneumococcal Polysaccharide (PnPs) Serotype 19A Antibody Response at 4 Weeks Postvaccination.
Description: GMT of the PnPs serotype 19A antibody response at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 and those who receive ZOSTAVAX™ and PNEUMOVAX™ 23 nonconcomitantly.
Time Frame: Four weeks postvaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/mL
Arm/Group | Nonconcomitant Group | Concomitant Group
Number analyzed (Participants) | 228 | 219
micrograms/mL | 10.5 [8.7 to 12.6] | 10.5 [8.7 to 12.7]
Statistical Analysis 1: Comparison: Nonconcomitant Group vs Concomitant Group; The hypothesis was that the GMT of the PnPs antibody responses to serotype 19A at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 will be noninferior to those in subjects who receive ZOSTAVAX™ nonconcomitantly; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, longitudinal regression model — The threshold for statistical significance is 0.025. There is no adjustment for multiple comparisons; [statistical method as in outcome 1, analysis 1]

7. Primary Outcome: Geometric Mean Titer (GMT) of the Pneumococcal Polysaccharide (PnPs) Serotype 22F Antibody Response at 4 Weeks Postvaccination.
Description: GMT of the PnPs serotype 22F antibody response at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 and those who receive ZOSTAVAX™ and PNEUMOVAX™ 23 nonconcomitantly.
Time Frame: Four weeks postvaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/mL
Arm/Group | Nonconcomitant Group | Concomitant Group
Number analyzed (Participants) | 228 | 219
micrograms/mL | 2.8 [2.3 to 3.3] | 2.5 [2.1 to 3.0]
Statistical Analysis 1: Comparison: Nonconcomitant Group vs Concomitant Group; The hypothesis was that the GMT of the PnPs antibody responses to serotype 22F at 4 weeks postvaccination in subjects who receive ZOSTAVAX™ concomitantly with PNEUMOVAX™ 23 will be noninferior to those in subjects who receive ZOSTAVAX™ nonconcomitantly; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, longitudinal regression model — The threshold for statistical significance is 0.025. There is no adjustment for multiple comparisons; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Nonconcomitant Group | Concomitant Group
Serious Adverse Events (participants affected / at risk) | 4 | 2
Other Adverse Events (participants affected / at risk) | 154 | 143
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Nonconcomitant Group | Concomitant Group
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0/236 | 1/235
Vertigo (Ear and labyrinth disorders) | 0/236 | 1/235
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/236 | 0/235
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/236 | 0/235
Haematoma (Vascular disorders) | 1/236 | 0/235
Diverticulitis (Infections and infestations) | 1/236 | 0/235
Global amnesia (Nervous system disorders) | 1/236 | 0/235
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Nonconcomitant Group | Concomitant Group
Nausea (Gastrointestinal disorders) | 3/236 | 2/235
Stomach discomfort (Gastrointestinal disorders) | 0/236 | 3/235
Vomiting (Gastrointestinal disorders) | 3/236 | 0/235
Fatigue (General disorders) | 3/236 | 1/235
Malaise (General disorders) | 0/236 | 3/235
Pyrexia (General disorders) | 1/236 | 5/235
Nasopharyngitis (Infections and infestations) | 5/236 | 9/235
Upper respiratory tract infection (Infections and infestations) | 1/236 | 5/235
Urinary tract infection (Infections and infestations) | 4/236 | 3/235
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/236 | 1/235
Back pain (Musculoskeletal and connective tissue disorders) | 5/236 | 3/235
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3/236 | 1/235
Myalgia (Musculoskeletal and connective tissue disorders) | 4/236 | 4/235
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4/236 | 2/235
Headache (Nervous system disorders) | 4/236 | 13/235
Cough (Respiratory, thoracic and mediastinal disorders) | 0/236 | 3/235
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4/236 | 5/235
Erythema (Skin and subcutaneous tissue disorders) | 3/236 | 3/235
Pruritus (Skin and subcutaneous tissue disorders) | 3/236 | 2/235
Rash (Skin and subcutaneous tissue disorders) | 6/236 | 1/235
Rash Vesicular (Skin and subcutaneous tissue disorders) | 4/236 | 3/235
Erythema (ZOSTAVAX™ injection site) (General disorders) | 70/236 | 72/235
Erythema (PNEUMOVAX™ 23 injection site) (General disorders) | 30/236 | 46/235
Erythema (Placebo injection site) (General disorders) | 7/236 | 1/235
Induration (ZOSTAVAX™ injection site) (General disorders) | 3/236 | 2/235
Pain (ZOSTAVAX™ injection site) (General disorders) | 68/236 | 74/235
Pain (PNEUMOVAX™ 23 injection site) (General disorders) | 82/236 | 95/235
Pain (Placebo injection site) (General disorders) | 21/236 | 8/235
Pruritus (ZOSTAVAX™ injection site) (General disorders) | 8/236 | 11/235
Swelling (ZOSTAVAX™ injection site) (General disorders) | 63/236 | 67/235
Swelling (PNEUMOVAX™ 23 injection site) (General disorders) | 30/236 | 49/235
Swelling (Placebo injection site) (General disorders) | 5/236 | 3/235

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.